CLINICAL TRIAL: NCT07376590
Title: Multicenter Study to Evaluate the Effectiveness and Safety of Flow-Diverting Stents for Distal Intracranial Aneurysms
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FESTR-DAN
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Aneurysms
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Device: Yes

INTERVENTIONS:
Device: No intervention measures — No intervention measures, Using data obtained from the treatment of intracranial distal intracranial aneurysms with flow diverter, evaluate the effecy and safety of blood flow diverter for the endovascular treatment of distal intracranial aneurysms.

SUMMARY:
Using data obtained from the treatment of intracranial distal intracranial aneurysms with flow diverter, evaluate the effecy and safety of blood flow diverter for the endovascular treatment of distal intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years, any gender，Subjects who have accepted treatment with flow-diverting for distal intracranial aneurysms
2. Diagnosed with an intracranial aneurysm by CTA, MRA, or DSA, with the following features: a wide neck (≥4mm), or a dome-to-neck ratio <2, saccular, fusiform aneurysms, recurrent saccular aneurysms, and dissecting aneurysms. Locations include: the Circle of Willis and it's distal branches such as the middle cerebral artery (MCA) M1-M3 segments, anterior cerebral artery (ACA) A1-A3 segments, posterior cerebral artery (PCA) P1-P2 segments, etc. (intracranial aneurysms of the Circle of Willis and it's distal vessels).
3. Subject or guardian is able to understand the purpose of study, shows sufficient compliance with the study protocol and provides a signed informed consent form

Exclusion Criteria:

1. Conditions that are not appropriate for stent delivery and deployment judged by investigators (severe stenosis of parent artery, severe tortuosity of parent artery, stent failing to reach the lesion, stent in the target lesion of parent artery, etc.)
2. mRS score ≥3
3. Heart, lung, liver and renal failure or other severe diseases (intracranial tumor, systemic infection, disseminated intravascular coagulation, myocardial infarction within 12 months before enrollment, history of severe psychosis, severe stenosis or occlusion of cerebral feeding artery, etc.)
4. Platelet count <60×10^9/L, known platelet dysfunction, or international normalized ratio (INR) >1.5
5. Major surgery within 30 days before enrollment，or planned to undergo surgery within 360 days after enrollment
6. Known allergies or contraindications to anesthetics, anticoagulants, and antiplatelet drugs
7. Pregnant or breastfeeding women
8. Subject has participated in other clinical trials within 1 month before signing informed consent
9. Other conditions judged by the investigators as unsuitable for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obtained from the treatment of intracranial distal intracranial aneurysms with flow diverter
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete occlusion rate of aneurysm 12 months after surgery | 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China